CLINICAL TRIAL: NCT02937740
Title: A 150-Day, Prospective, Phase 4, Open-Label Study, Evaluating Patient Satisfaction and Symptom Improvement When Treating Male Hypogonadism With Testosterone Nasal Gel (Natesto™)
Brief Title: Open-Label Study, Evaluating Patient Satisfaction and Symptom Improvement When Treating Male Hypogonadism With Natesto™
Acronym: MyT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Acerus Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAT-2016-01
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Results first posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-07

CONDITIONS: Hypogonadism
Keywords: Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Natesto

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naive patients - ARM 1 (Other): NATESTO Testosterone Nasal Gel administered intranasally to patients with no prior TRT experience. Multiple-dose dispenser will be used for gel deposition into the nasal cavity. The dispenser is a finger-actuated, non-pressurized dispensing system designed to deliver 122.5mg of NATESTO (5.5mg testosterone) per actuation.
  For BID administration, NATESTO 22 mg/day of testosterone. For the subset of patients that continue on TID, NATESTO 33 mg/day of testosterone.
  Interventions: Drug: NATESTO Testosterone Nasal Gel
- Non-naive patients - ARM 2 (Other): NATESTO Testosterone Nasal Gel administered intranasally to patients who had prior TRT. Multiple-dose dispenser will be used for gel deposition into the nasal cavity. The dispenser is a finger-actuated, non-pressurized dispensing system designed to deliver 122.5mg of NATESTO (5.5mg testosterone) per actuation.
  For BID administration, NATESTO 22 mg/day of testosterone. For the subset of patients that continue on TID, NATESTO 33 mg/day of testosterone.
  Interventions: Drug: NATESTO Testosterone Nasal Gel

INTERVENTIONS:
Drug: NATESTO Testosterone Nasal Gel — Participants will be instructed to administer 5.5 mg of testosterone (1 actuation) per nostril of NATESTO Testosterone Nasal Gel once in the morning and once in the evening (at least 6 hours apart), preferably at the same time each day for a total daily dose of 22 mg/day of testosterone. Patients should be instructed to completely depress the pump 1 time in each nostril to receive the total dose.
  For three times daily (after Visit 4 [Day 90] if symptoms not adequately managed by a BID dose), NATESTO will be administered intranasally once in the morning, once in the afternoon and once in the evening (approximately 6-8 hours apart), preferably at the same time each day for a total daily dose of 33 mg/day of testosterone.
  Other Names: NATESTO

SUMMARY:
Multicenter study consisting of two study periods as follows: a 90-day Treatment Period, with potential extension by 30 days for those patients requiring a dose increase, as determined by the treating physician. Participants receiving 122.5mg of NATESTO (5.5 mg of testosterone) per nostril twice daily may have an increased daily dose adjustment on Day 90, based on their hypogonadism symptoms.

DETAILED DESCRIPTION:
The primary objective of the study is to measure patient satisfaction with testosterone replacement therapy before (for non-naïve patients), during and after treatment with NATESTO.

The secondary objectives of this study are to evaluate the following:

* Improvement in hypogonadism symptoms;
* Patient treatment preference versus prior testosterone replacement therapy;
* Frequency of daily dose of NATESTO;
* Safety monitoring.

The population for this study is adult men 18-65 years of age inclusive, with primary or secondary hypogonadism, with historical documented total serum testosterone concentration of ≤300 ng/dL and the ability to provide informed consent. Eligible subjects include treatment-naïve, hypogonadal patients with a documented confirmation of hypogonadism, as well as patients previously treated with an alternate topical testosterone replacement therapy (TRT) for at least three months prior to selection. Participants currently receiving topical testosterone replacement therapy will be required to discontinue their current testosterone treatment before initiating treatment with NATESTO. The approximate total duration of study participation for participants completing the study will be up to 150 days (~21 weeks).

This is a Phase 4, multicenter study consisting of two study periods as follows:

* A 90-day Treatment Period, extended to 120-days for those subjects requiring a dose increase, during which participants will receive 122.5 mg of NATESTO (5.5mg testosterone) per nostril twice daily (BID) for 90 days. At Day 90, the treating physician will assess the patient's hypogonadism symptoms, review patient's completed questionnaires and based on the Canadian Men's Health Foundation Multidisciplinary Guidelines as endorsed by both the Canadian Urological Association and the Canadian Society of Endocrinology and Metabolism1, decide if continuation at a higher dose frequency of three-times daily (TID) is required for efficacy. For TID patients, there will be a 30-day Treatment Extension during which participants whose symptoms were not adequately treated on a BID dose, will receive 122.5 mg of NATESTO TID (5.5mg testosterone) per nostril. At Day 120, the TID patient will return to the site for examination, discussion of symptoms with the physician and questionnaire completion. All patients will have their blood testosterone levels assessed at Day 90 and only TID patients at Day 120.
* Post-study follow-up: All study patients will be requested to follow up at Day 150 to confirm whether they continued therapy with NATESTO.

Patient selection will come as a result of a doctor's visit for routine controls, prescription renewal and by pre-selection by the physician from among hypogonadal patients currently receiving topical testosterone replacement therapies and willing to participate in a clinical trial with NATESTO, or as a result of an initial consultation for naïve patients.

At Visit 1, patients who agree to participate in the study will come to the site. They will provide written informed consent and undergo a complete physical examination, including a nasal examination, and medical history collection. Blood pressure, heart rate, weight, and height measurements (from which body mass index [BMI] will be determined) will also be performed. Blood will be drawn at a local lab for safety assessment. However, if these values have already been documented in their patient file from the preceding 6 months, then those values will be entered into the eCRF. Previous treatment for hypogonadism (drug and nondrug; daily dose) will be recorded, as well as other concomitant treatment with drug or nondrug therapies. Study questionnaires Treatment Satisfaction Questionnaire for Medication (TSQM) and quantitative Androgen Deficiency in the Aging Male (qADAM) will be reviewed and subjects will be given instructions for proper completion of the instruments. Patients will complete Part A of the Patient Preference and Use Questionnaire. Patients will also be provided with a prescription for a 90-day supply of the study medication, NATESTO, and a Study Drug Access Card that will be used for payment purposes at the patient's preferred pharmacy.

Non-naïve participants will be instructed to stop their current topical treatment at least one day and no more than 7 days prior to initiation of treatment with NATESTO. Patients should not take both medications simultaneously.

The open-label Treatment Period will consist of a maximum of 5 study visits: 2 visits will be done via telephone by the Study Coordinator (Visit 2, Day 30 and Visit 3, Day 60) and one clinic visit (Visit 4, Day 90), and a last clinic visit for patients who were placed on a TID dose (Visit 5, Day 120).

At Visit 2 (Day 30) and Visit 3 (Day 60), participants will be required to complete questionnaires (TSQM and qADAM) by telephone with the Study Coordinator, and will also be asked about any concurrent medications or AEs.

At Visit 4 (Day 90), the patient will return to the site. Any unreported adverse events will be recorded. Patients will undergo a basic physical examination including a nasal examination. Blood pressure, heart rate, weight, and height measurements (from which body mass index [BMI] will be determined) will be recorded. Hypogonadism symptoms will be assessed by the Investigator making reference to the qADAM questionnaire results, and the patient will complete the TSQM.

At Visit 4 (Day 90), if in the physician's judgment the patient is adequately treated with twice daily (BID) NATESTO, the physician will decide whether the patient a.) should return to their previous therapy; b.) remain on NATESTO; or c.) consider a new treatment option. The physician will provide the patient with a prescription for the treatment chosen. The BID patients will have a blood draw taken at a local laboratory for safety assessment and to assess their testosterone level. This will constitute the END OF TREATMENT for BID subjects. These adequately controlled patients will complete Part B (for Non-naïve) or Part C (for Naïve) of the Patient Preference and Use Questionnaire.

At Visit 4 (Day 90), if the physician's judgement is that the twice daily (BID) dose of NATESTO was not adequate to treat the patient's symptoms and believes that the patient will benefit from a higher dose, then a prescription will be given to the patient for three times daily (TID) NATESTO. The Study Drug Access Card will be used for payment purposes at the patient's preferred pharmacy. These patients moving to TID will have a blood draw taken at a local laboratory to assess safety as well as their testosterone level. The patient will schedule Visit 5 (Day 120) at this time.

At Visit 5 (Day 120 for TID patients only), any unreported adverse events will be recorded. Patients will undergo a basic physical examination including a nasal examination. Blood pressure, heart rate, weight, and height measurements (from which body mass index [BMI] will be determined) will be recorded. The patients will have a blood draw taken at a local laboratory for safety assessment and to assess their testosterone level. In addition to TSQM and qADAM questionnaires, subjects will also complete Part B (for Non-naïve) or Part C (for Naïve) of the Patient Preference and Use Questionnaire. The physician will decide whether the patient a.) should return to their previous therapy; b.) remain on NATESTO; or c.) consider a new treatment option. The physician will provide the patient with a prescription for the treatment chosen.

At Visit 6 (Day 150), all study patients will be asked by telephone whether they are still taking NATESTO and why (or why not).

ELIGIBILITY:
Inclusion Criteria:

* Hypogonadal male between 18 and 65 years of age, inclusive;
* Able to understand and provide signed informed consent;
* Have documented total serum testosterone levels ≤300 ng/dL;
* Are currently being treated with any form of a topical testosterone replacement therapy for at least three months, or are treatment-naive.

Exclusion Criteria:

* In the opinion of the Investigator, significant intercurrent disease of any type, in particular liver, kidney, heart disease, stroke, or psychiatric illness;
* History of pituitary or hypothalamic tumors or history of any malignancy (including breast and prostate cancers) excluding basal cell or squamous cell carcinoma of the skin curatively treated by surgery;
* Prostatomegaly or history of abnormal PSA levels (>10.0 ng/mL). If PSA is >10 ng/mL, a recent negative biopsy must be documented (within the last 12 months);
* History of nasal disorders, nasal or sinus surgery, nasal fracture within the previous 6 months or nasal fracture that caused a deviated anterior nasal septum surgery, mucosal inflammatory disorders, specifically Sjogren's syndrome;
* Use of any form of intranasal medication delivery other than periodic short-term (less than 3 days) use of sympathomimetic decongestants;
* History of severe adverse drug reactions to testosterone therapies;
* History or current evidence of abuse of alcohol or any drug substance;
* Current treatment with other androgens (e.g., dehydroepiandrosterone [DHEA]), anabolic steroids, or other sex hormones;
* Treatment with estrogens, gonadotropin-releasing hormone (GnRH) agonists, or growth hormone within the previous 12 months;
* Treatment with drugs that interfere with the metabolism of testosterone, such as anastrozole, clomiphene, dutasteride, finasteride, flutamide, ketoconazole, spironolactone, or testolactone;
* Poor compliance history;
* Participation in any other research study during the conduct of this study or 30 days prior to the initiation of this study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2016-10; Primary Completion 2017-10 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Bryson, Ph.D., Study Director — Sponsor GmbH
Locations (11):
- Canada (11):
  - Prostate Cancer Centre - Research, Calgary, Alberta
  - Silverado Research Inc., Victoria, British Columbia
  - LMC Barrie, Barrie, Ontario
  - G. Kenneth Jansz Medicine Professional Corporation, Burlington, Ontario
  - Lawson Research Institute / St Joseph's Health Care London, London, Ontario
  - The Fe/Male Health Centre, Oakville, Ontario
  - Toronto Urology Clinical Study Group, Toronto, Ontario
  - Rabih Nour Clinic Windsor, Windsor, Ontario
  - Ultra-Med Inc., Pointe-Claire, Quebec
  - Clinique D'Andropause de Quebec, Québec, Quebec
  - Dr. Carlos Marois Urologue, Verdun, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Naive Patients - ARM 1: NATESTO Testosterone Nasal Gel administered intranasally to patients with no prior TRT experience. Multiple-dose dispenser will be used for gel deposition into the nasal cavity. The dispenser is a finger-actuated, non-pressurized dispensing system designed to deliver 122.5mg of NATESTO (5.5mg testosterone) per actuation.
  For BID administration, NATESTO 22 mg/day of testosterone. For the subset of patients that continue on TID, NATESTO 33 mg/day of testosterone.
  NATESTO Testosterone Nasal Gel: Participants will be instructed to administer 5.5 mg of testosterone (1 actuation) per nostril of NATESTO Testosterone Nasal Gel once in the morning and once in the evening (at least 6 hours apart), preferably at the same time each day for a total daily dose of 22 mg/day of testosterone. Patients should be instructed to completely depress the pump 1 time in each nostril to receive the total dose.
  For three times daily (after Visit 4 [Day 90] if symptoms not adequately managed by a BID
- Non-naive Patients - ARM 2: NATESTO Testosterone Nasal Gel administered intranasally to patients who had prior TRT. Multiple-dose dispenser will be used for gel deposition into the nasal cavity. The dispenser is a finger-actuated, non-pressurized dispensing system designed to deliver 122.5mg of NATESTO (5.5mg testosterone) per actuation.
  For BID administration, NATESTO 22 mg/day of testosterone. For the subset of patients that continue on TID, NATESTO 33 mg/day of testosterone.
  NATESTO Testosterone Nasal Gel: Participants will be instructed to administer 5.5 mg of testosterone (1 actuation) per nostril of NATESTO Testosterone Nasal Gel once in the morning and once in the evening (at least 6 hours apart), preferably at the same time each day for a total daily dose of 22 mg/day of testosterone. Patients should be instructed to completely depress the pump 1 time in each nostril to receive the total dose.
  For three times daily (after Visit 4 [Day 90] if symptoms not adequately managed by a BID dose), NATE
Period: BID for 90 Days, 22 mg/Day
Arm/Group | Naive Patients - ARM 1 | Non-naive Patients - ARM 2
Started | 24 | 93
Completed | 19 | 62
Not Completed | 5 | 31
Not completed — Withdrawal by Subject | 3 | 14
Not completed — Adverse Event | 0 | 10
Not completed — Lost to Follow-up | 2 | 7
Period: Uptitrated to TID on Day 90 for 30 Days
Arm/Group | Naive Patients - ARM 1 | Non-naive Patients - ARM 2
Started | 13 | 17
Completed | 12 | 15
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Missed visits | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Naive Patients - ARM 1: NATESTO Testosterone Nasal Gel administered intranasally to patients with no prior TRT experience. Multiple-dose dispenser will be used for gel deposition into the nasal cavity. The dispenser is a finger-actuated, non-pressurized dispensing system designed to deliver 5.5mg testosterone per actuation.
  For BID administration, NATESTO 22 mg/day of testosterone. For the subset of patients that continue on TID, NATESTO 33 mg/day of testosterone.
  To be given three times daily (after Visit 4 [Day 90]) if symptoms not adequately managed on BID.
- Non-naive Patients - ARM 2: NATESTO Testosterone Nasal Gel administered intranasally to patients who had prior TRT. Multiple-dose dispenser will be used for gel deposition into the nasal cavity. The dispenser is a finger-actuated, non-pressurized dispensing system designed to deliver 5.5mg testosterone per actuation.
  For BID administration, NATESTO 22 mg/day of testosterone. For the subset of patients that continue on TID, NATESTO 33 mg/day of testosterone.
  To be given three times daily (after Visit 4 [Day 90]) if symptoms not adequately managed on BID.
- Total: Total of all reporting groups
Arm/Group | Naive Patients - ARM 1 | Non-naive Patients - ARM 2 | Total
Number analyzed (Participants) | 23 | 77 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (11.6) | 52.9 (8.2) | 52.8 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 23 | 77 | 100
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 8 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 20 | 68 | 88
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction - Change From Baseline
Description: The primary objective of this study is to measure patient satisfaction with testosterone replacement therapy before, during and after treatment with NATESTO. Patient satisfaction with treatment will be measured by TSQM (Treatment Satisfaction Questionnaire for Medication) Version 9, a 9-item validated instrument. TSQM domains include - Effectiveness, Convenience, Global Satisfaction. The score for each domain is converted into a scale out of 100. Higher values imply a better outcome.
Time Frame: Baseline and 3 months for BID, 4 months for TID
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Natesto Testosterone Intranasal Gel Given BID: Patients who completed 90 days on BID NATESTO.
- Natesto Testosterone Intranasal Gel Given TID: Patients who completed 90 days on BID NATESTO and were then switched to TID treatment for an additional 30 days.
Arm/Group | Natesto Testosterone Intranasal Gel Given BID | Natesto Testosterone Intranasal Gel Given TID
Number analyzed (Participants) | 47 | 15
Units on a scale
  Effectiveness Domain Change from Baseline | 9.6 (25.9) | 21.5 (14.4)
  Convenience Domain Change from Baseline | 18.9 (21.4) | 21.9 (24.8)
  Global Satisfaction Domain Change from Baseline | -0.6 (33.0) | 13.3 (22.9)

2. Secondary Outcome: Change in Hypogonadism Symptoms
Description: Change in hypogonadism symptoms from baseline as measured by qADAM, a 10 point validated instrument. qADAM is a 10-item, patient-reported outcome measure used to evaluate the symptom severity of hypogonadism. Responses can range from 1 to 5 per question allowing for a minimum to maximum score range of 10 to 50. Higher values imply a better outcome.
Time Frame: Baseline and 3 months for BID, 4 months for TID
Population: ITT population, no-LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Non-naive Patients - BID Treatment: NATESTO Testosterone Nasal Gel administered intranasally to patients who had prior TRT.
  For BID administration, NATESTO 22 mg/day of testosterone. Change in scores is between Day 90 and Baseline.
- Naive Patients - BID Treatment: NATESTO Testosterone Nasal Gel administered intranasally to patients with no prior TRT experience.
  For BID administration, NATESTO 22 mg/day of testosterone. Change in scores is between Day 90 and Baseline.
- Non-naive Patients - TID Treatment: NATESTO Testosterone Nasal Gel administered intranasally to patients previously on TRT.
  Patients whose symptoms were not adequately controlled on BID treatment at Study Day 90 were switched to TID (33 mg/day) for 30 days. Change in scores is between Day 120 and Baseline.
- Naive Patients - TID Treatment: NATESTO Testosterone Nasal Gel administered intranasally to patients with no prior TRT experience.
  Patients whose symptoms were not adequately controlled on BID treatment at Study Day 90 were switched to TID (33 mg/day) for 30 days. Change in scores is between Day 120 and Baseline.
Arm/Group | Non-naive Patients - BID Treatment | Naive Patients - BID Treatment | Non-naive Patients - TID Treatment | Naive Patients - TID Treatment
Number analyzed (Participants) | 47 | 7 | 15 | 12
Units on a scale | 4.8 (6.5) | 12.0 (3.9) | 3.9 (3.8) | 6.8 (4.1)

3. Secondary Outcome: Patient Treatment Preference Versus Prior Testosterone Replacement Therapy
Description: Patient treatment preference versus prior testosterone replacement therapy measured by the Treatment Preference questionnaire.
Time Frame: Last visit, i.e. 3 months for BID, 4 months for TID
Population: Number of participants includes BID and TID patients for each Arm. The number is different than the total number of patients who completed because some subjects did not provide a response to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Naive Patients - ARM 1 | Non-naive Patients - ARM 2
Number analyzed (Participants) | 18 | 54
Participants
  Yes, I plan to continue taking NATESTO | 10 | 32
  I am undecided if I will continue NATESTO | 5 | 12
  No, I do not plan to continue taking NATESTO | 3 | 10

4. Secondary Outcome: Frequency of Daily Dose of NATESTO by the End of the Study
Description: Frequency of daily dosing, i.e. how many patients remained on BID vs how many were uptitrated to TID by the end of the study.
Time Frame: 3 months for those who remained on BID, 4 months for those uptitrated to TID
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Naive Patients - ARM 1 | Non-naive Patients - ARM 2
Number analyzed (Participants) | 23 | 77
Participants
  BID | 10 | 60
  TID | 13 | 17

ADVERSE EVENTS:
Time Frame: 90 or 120 days
Arm/Group | Natesto Testosterone Intranasal Gel Given BID | Natesto Testosterone Intranasal Gel Given TID
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/87 | 0/30
Other Adverse Events (participants affected / at risk) | 22/87 | 5/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Natesto Testosterone Intranasal Gel Given BID (N=87) | Natesto Testosterone Intranasal Gel Given TID (N=30)
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Natesto Testosterone Intranasal Gel Given BID (N=87) | Natesto Testosterone Intranasal Gel Given TID (N=30)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dysgeusia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Epistaxis (Vascular disorders) | 5 (5) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-02-13): https://cdn.clinicaltrials.gov/large-docs/40/NCT02937740/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/40/NCT02937740/SAP_001.pdf